CLINICAL TRIAL: NCT06990178
Title: Adaptive Neoadjuvant Therapy for Esophageal Cancer:A Multicenter Phase II Clinical Trail
Brief Title: Adaptive Neoadjuvant Therapy for Esophageal Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other)
Responsible Party: Principal Investigator, Wei Jiang, Associate chief physician, Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eso2025510
Record Dates: First submitted 2025-05-11; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Carcinoma; Neoadjuvant Therapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a multicenter, single-arm, phase II study. The purpose of this study is to evaluate the efficacy and safety of adaptive neoadjuvant therapy combining neoadjuvant chemotherapy and immunotherapy with concurrent low-dose radiotherapy ± chemoradiotherapy in treatment-naive patients with resectable esophageal squamous cell carcinoma (ESCC) at stages T1-4aN1-3M0 or T3-4aN0M0.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemotherapy + immunotherapy+ low-dose radiotherapy (4Gy/2F) (Experimental): Eligible ESCC patients will receive standard neoadjuvant chemotherapy + immunotherapy, low-dose radiotherapy (4Gy/2F), and chemotherapy + immunotherapy (regimen: albumin-bound paclitaxel + carboplatin + tislelizumab q3w). After two cycles, imaging and endoscopic ultrasound, as well as pathological evaluations will be conducted. Patients will be stratified based on whether they achieve complete clinical response (cCR). The cCR group will undergo radical surgery, while the non-cCR group will continue with neoadjuvant concurrent chemoradiotherapy (2Gy*20f) followed by radical surgery. Postoperative adjuvant therapy will be administered as per routine
  Interventions: Radiation: Neoadjuvant concurrent chemoradiotherapy

INTERVENTIONS:
Radiation: Neoadjuvant concurrent chemoradiotherapy — Non-cCR group will continue with neoadjuvant concurrent chemoradiotherapy (2Gy*20f) followed by radical surgery

SUMMARY:
This study is a multicenter, single-arm phase II trial, aiming to evaluate the efficacy and safety of neoadjuvant chemotherapy and immunotherapy combined with concurrent low-dose radiotherapy ± chemoradiotherapy as an adaptive neoadjuvant treatment for previously untreated resectable esophageal squamous cell carcinoma. Compared with neoadjuvant concurrent chemoradiotherapy, the pathological complete response (pCR) rate of neoadjuvant chemoradiotherapy is lower, and non-pCR has a relatively poorer prognosis than pCR. Therefore, how to further increase the pCR rate of neoadjuvant chemoradiotherapy under the premise of minimum toxicity is an important link to improve the efficacy of this treatment strategy. Low-dose radiotherapy provides an option for this strategy. Compared with traditional high-dose radiotherapy, low-dose radiotherapy is very safe, and the extremely low radiotherapy dose causes almost negligible damage to normal tissues. However, it can effectively reshape the immune microenvironment, converting cold tumors into hot tumors. On this basis, combined with immune checkpoint inhibitors, it can achieve effective immune responses in advanced tumors, bringing new hope for the treatment of advanced tumor patients. Low-dose radiotherapy can regulate the tumor immune microenvironment through multiple mechanisms and enhance the body's anti-tumor immune response, thus potentially further improving the efficacy of neoadjuvant chemoradiotherapy for esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for esophageal cancer:

1. Histologically or cytologically confirmed thoracic esophageal squamous cell carcinoma (ESCC) at stages T1-4aN1-3M0 or T3-4aN0M0 (AJCC 9th edition); Neck color Doppler ultrasound shows no suspicious metastatic lymph nodes.

   Note: For the determination of T staging, CT combined with MRI or endoscopic ultrasound is used. Research centers are encouraged to use endoscopic ultrasound; Research centers are encouraged to obtain tissue confirmation of lymph node involvement, provided that it can be safely obtained through puncture, EBUS (endobronchial ultrasound), EUS (endoscopic ultrasound) or mediastinoscopy. However, when the boundaries of the lymph nodes are clear and the shortest axis diameter of at least one lymph node is ≥ 2.0 cm, lymph node involvement can be determined by imaging examination (MRI/CT scan); M1 is excluded in FDG-PET/CT or diagnostic-quality CT or MRI scans of the chest, abdomen, pelvis and brain.
2. The lesion is a potentially resectable thoracic esophageal lesion.
3. R0 resection is expected to be achieved.
4. No previous treatment for esophageal tumors has been received.

General inclusion requirements:

1. Sign the informed consent form.
2. Male or female aged ≥ 18 years and ≤ 75 years.
3. ECOG performance status is 0 or 1.
4. There are no surgical contraindications based on the evaluation of various organ function tests before surgery.
5. Body weight is greater than 35 kg; The weight loss in the past three months does not exceed 10%.
6. The expected survival time is more than 12 months.
7. Agree to provide previously stored tumor tissue specimens or undergo a biopsy to collect tumor lesion tissue for biomarker analysis.
8. According to the RECIST 1.1 criteria, there is at least one measurable lesion.
9. Good organ function:

A.Hematology:

White blood cell count ≥ 4×10⁹/L Neutrophil count ≥ 2×10⁹/L Hemoglobin ≥ 9 g/dL Platelet count ≥ 100×10⁹/L

B.Liver function:

Bilirubin ≤ 1.5 times the upper limit of normal (ULN). Patients with known Gilbert's disease and a serum bilirubin level ≤ 3 times ULN may be eligible for enrollment.

Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN. In case of liver metastasis, AST/ALT ≤ 5 times ULN.

Alkaline phosphatase (ALP) ≤ 3 times ULN. In case of liver or bone metastasis, ALP ≤ 5 times ULN.

Albumin ≥ 3 g/dL International Normalized Ratio (INR), Prothrombin Time (PT) or Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 times ULN

C.Renal function:

Serum creatinine ≤ 1.5 times ULN or creatinine clearance rate ≥ 60 mL/min calculated by the Cockcroft - Gault formula

Exclusion Criteria:

Cancer - specific exclusion criteria:

1. Cervical esophageal cancer. Patients whose clinical stage is determined to be stage I/IIA, unresectable stage T4b, or with distant metastasis (M1) through imaging examinations such as enhanced chest - abdomen CT, cervical lymph node ultrasound, whole - body PET - CT, or EBUS (optional).
2. Patients with a history of malignancies other than esophageal cancer within 5 years, except for malignancies with negligible risk of metastasis or death (e.g., expected 5 - year overall survival rate > 90%) and those expected to be cured after treatment, such as appropriately treated cervical carcinoma in situ, basal or squamous cell skin cancer, limited prostate cancer treated with radical surgery, and ductal carcinoma in situ treated with radical surgery.

General medical exclusion criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the study period.
2. Patients with a history of idiopathic pulmonary fibrosis, organizing pneumonia (such as bronchiolitis obliterans), drug - induced pneumonia, idiopathic pneumonia, or evidence of active pneumonia detected by chest CT scan during screening.
3. Significant cardiovascular diseases, such as heart diseases defined by the New York Heart Association (class II or higher), myocardial infarction occurring within 3 months before enrollment, unstable arrhythmia, unstable angina pectoris. Patients known to have coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must receive the optimal stable treatment plan determined by the attending physician, and consultation with a cardiologist can be carried out if necessary.
4. Patients with active hepatitis B (chronic or acute; defined as positive hepatitis B surface antigen (HBsAg) test result during screening and HBV DNA copy number > 1000 cps/ml) or hepatitis C:
5. Patients with a history of hepatitis B virus (HBV) infection or those with cured HBV infection (defined as positive hepatitis B core antibody (HBcAb) and negative HBsAg) may be eligible for this study. Before random assignment, HBV deoxyribonucleic acid (DNA) testing must be performed on such patients, and they are only eligible to participate in the study if HBV DNA is negative (HBV DNA < 1000 cps/ml).
6. Among patients with positive hepatitis C virus (HCV) antibody, only those with negative polymerase chain reaction (PCR) HCV ribonucleic acid (RNA) can participate in this study.
7. Patients with active pulmonary tuberculosis (clinical diagnosis includes clinical history, physical examination, imaging findings, and TB examinations according to local medical routines).
8. Patients with a positive human immunodeficiency virus (HIV) test result.
9. Patients with severe uncontrolled systemic intermittent diseases, such as active infections or poorly controlled diabetes.
10. Patients with abnormal blood coagulation function, bleeding tendency (such as active peptic ulcer), or those receiving thrombolytic or anticoagulant therapy.
11. Patients with existing or co - existing hemorrhagic diseases.
12. Patients with peripheral nervous system disorders or a history of significant mental disorders and central nervous system disorders.
13. Patients who, due to previous surgeries, cannot use the stomach to replace the esophagus for digestive tract reconstruction in this surgery.

Treatment - related exclusion criteria:

1. Patients who have received any approved anti - cancer treatment (including radiotherapy, chemotherapy, hormone therapy, or traditional Chinese medicine) before starting the study treatment.
2. Patients who have received other investigational drugs or participated in other therapeutic clinical studies within 28 days before enrollment; this includes signing the informed consent form (ICF) for other trials, and patients who failed screening are also not eligible for enrollment.
3. Patients who have previously received immune checkpoint blockade therapy, such as treatment with anti - programmed death receptor - 1 (anti - PD - 1) and anti - PD - L1 therapeutic antibodies.
4. Patients who have received systemic immunostimulants within 4 weeks before random assignment or within 5 drug half - lives (t1/2) (whichever is longer) [including but not limited to interferon (IFN) or interleukin - 2]; vaccination with cancer vaccines is allowed in previous treatments.
5. Patients who have received systemic immunosuppressive drugs (> 10 mg/d prednisone equivalent) within 2 weeks before random assignment, including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti - tumor necrosis factor (TNF) drugs:
6. For patients who have received short - term, low - dose, systemic immunosuppressive treatment (for example, a single dose of dexamethasone for nausea), they may participate in this study after consultation between the investigator and the medical monitor and approval by the medical monitor.
7. Patients using inhaled corticosteroids for the treatment of chronic obstructive pulmonary disease, patients using mineralocorticoids (such as fludrocortisone) for the treatment of orthostatic hypotension, and patients using low - dose glucocorticoid supplements (≤10mg /d prednisone or equivalent) for the treatment of adrenal cortical insufficiency are eligible for enrollment.
8. Patients with a history of allergic reactions to platinum - containing compounds or taxanes.
9. Other situations determined by the principal investigator (PI) or attending physician as inappropriate for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2028-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
pCR | Immediately after the surgery
  Pathological complete response rate

SECONDARY OUTCOMES:
EFS | 2 year
  EFS is defined as the time from randomization to the occurrence of disease progression or the time of death due to any cause (whichever occurs first), and it is determined by the Independent Review Committee (BIRC) according to the criteria.
ORR | Before surgery
OS | 2 year
R0 | Immediately after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhen Yu, MD, Principal Investigator — National Cancer Center/ Cancer Hospital &Shenzhen Hospital Chinese Academy of Medical Sciences and Peking Union Medical College; Wei Jiang, MD, Principal Investigator — National Cancer Center/ Cancer Hospital &Shenzhen Hospital Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- 113 Baohe Road,Longgang District,Shenzhen,China, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code